CLINICAL TRIAL: NCT04804020
Title: The Effectiveness and Safety of the Three Endometrial Preparation Protocols for Frozen Embryo Transfer Natural Cycle, Modified Natural Cycle and Artificial Cycle: a Randomized Controlled Trial
Brief Title: Natural Cycle vs. Modified Natural Cycle vs. Artificial Cycle Protocol for Endometrial Preparation.
Acronym: MONART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mỹ Đức Hospital (Other)
Collaborators: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 187/HĐĐĐ-ĐHYD
Record Dates: First submitted 2021-03-11; First posted 2021-03-18 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: IVF; Frozen Embryo Transfer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NC (Natural cycle) (Active Comparator): Performing the first ultrasound scan will be performed on the second to the fourth day of the menstrual cycle to identify any problem related to the patients' uterus or adnexa. The second ultrasound will be performed on the sixth day of the cycle. Daily ultrasound and serum estradiol and LH level evaluation will be performed when the mean diameter of the dominant follicle of ≥14 mm. LH surge initiation is defined as a concentration of 180% above the latest serum value available in that patient with a continued rise thereafter to a level of 20 IU/l or more detected by the ECLIA method (Roche Cobas® E 801, Roche Diagnostics, Germany). Embryo transfer will be scheduled by the time of the initiation of LH and embryo stages.
  Interventions: Procedure: NC
- mMC (modified Natural cycle) (Active Comparator): Performing the first ultrasound scan on the second to the fourth day of the menstrual cycle to identify any problem related to patients' uterus or adnexa. A second ultrasound scan will be performed on the sixth day of the cycle; if there is at least one follicle with a diameter of ≥12 mm, an ultrasound scan will be performed daily. When the dominant follicle's mean diameter is ≥16 mm, human chorionic gonadotropin (Ovitrelle® 250 μg; Merck, Kenilworth, NJ, USA) will be injected to trigger ovulation. Embryo transfer will be scheduled by the time of the hCG injection and embryo stages.
  Interventions: Procedure: mNC
- AC (Artificial cycle) (Active Comparator): Preparing the endometrium by using oral estradiol valerate (Valiera®; Laboratories Recalcine) 8 mg/day, ranging from the second or fourth menstruation day. The endometrial thickness will be monitored from day six onwards, and vaginal progesterone (Utrogestan®; Besins) 800 mg/day will be initiated when endometrial thickness reaches ≥7 mm. Estradiol exposure must be lasting for ≥9 days before progesterone administration. Embryo transfer will be scheduled by the time of the initiation of progesterone and embryo stages.
  Interventions: Procedure: AC

INTERVENTIONS:
Procedure: NC — The first ultrasound scan will be performed on the second to the fourth day of the menstrual cycle to identify any problem related to the patients' uterus or adnexa. The second ultrasound will be performed on the sixth day of the cycle. Daily ultrasound and serum estradiol and LH level evaluation will be performed when the mean diameter of the dominant follicle of ≥14 mm. LH surge initiation is defined as a concentration of 180% above the latest serum value available in that patient with a continued rise thereafter9 to a level of 20 IU/l or more10 detected by the ECLIA method (Roche Cobas® E 801, Roche Diagnostics, Germany). Embryo transfer will be scheduled by the time of the initiation of LH and embryo stages.
  Arms: NC (Natural cycle)
Procedure: mNC — The first ultrasound scan will be performed on the second to the fourth day of the menstrual cycle to identify any problem related to patients' uterus or adnexa. A second ultrasound scan will be performed on the sixth day of the cycle; if there is at least one follicle with a diameter of ≥12 mm, an ultrasound scan will be performed daily. When the dominant follicle's mean diameter is ≥16 mm, human chorionic gonadotropin (Ovitrelle® 250 μg; Merck, Kenilworth, NJ, USA) will be injected to trigger ovulation. Embryo transfer will be scheduled by the time of the hCG injection and embryo stages.
  Arms: mMC (modified Natural cycle)
Procedure: AC — The endometrium is prepared using oral estradiol valerate (Valiera®; Laboratories Recalcine) 8 mg/day, ranging from the second or fourth menstruation day. The endometrial thickness will be monitored from day six onwards, and vaginal progesterone (Utrogestan®; Besins) 800 mg/day will be initiated when endometrial thickness reaches ≥7 mm. Estradiol exposure must be lasting for ≥9 days before progesterone administration. Embryo transfer will be scheduled by the time of the initiation of progesterone and embryo stages.
  Arms: AC (Artificial cycle)

SUMMARY:
Fresh embryo transfer is a routine procedure in vitro fertilization (IVF) treatment. Since the first live birth after an IVF-FET (frozen embryo transfer), recent years have seen a dramatic rise in the number of FET cycles. Three endometrial preparation protocols for frozen-thawed embryo transfer, including artificial, natural, modified natural protocol, have been studied and applied to maximize treatment outcomes. However, those methods are being applied empirically as their efficacy and safety are yet to be determined. The objective of this study is to compare the effectiveness and safety of those protocols.

DETAILED DESCRIPTION:
This trial will be conducted at My Duc Hospital, Ho Chi Minh City, Viet Nam. Women who are potentially eligible will be provided information about the trial as long as their stimulation cycles are initiated. Screening for eligibility will be performed by treating physicians on day 2 of the menstrual cycle in the subsequent frozen embryo transfer cycles. Patients will be provided a copy of the informed consent documents. Written informed consent will be obtained by the investigator from all women before the enrolment. Women will be randomized (1:1:1) to AC (artificial cycle) or NC (natural cycle), or mNC (modified natural cycle) protocols using block randomization with a variable block size of 6 or 9 by an independent study coordinator via telephone, using a computer-generated random list (block size of 6, or 9).

Artificial protocol The endometrium is prepared using oral estradiol valerate (Valiera®; Laboratories Recalcine) 8 mg/day, ranging from the second or fourth menstruation day. The endometrial thickness will be monitored from day six onwards, and vaginal progesterone (Utrogestan®; Besins) 800 mg/day will be initiated when endometrial thickness reaches ≥7 mm. Estradiol exposure must be lasting for ≥9 days before progesterone administration. Embryo transfer will be scheduled by the time of the initiation of progesterone and embryo stages. In cases where a dominant follicle emerged, serum LH and progesterone will be determined to rule out luteinization. If LH concentrations are <13 IU and progesterone levels <15 nmol/l, luteinization will deem not to have occurred, and FET was performed.

Natural protocol The first ultrasound scan will be performed on the second to the fourth day of the menstrual cycle to identify any problem related to the patient's uterus or adnexa. The second ultrasound will be performed on the sixth day of the cycle. Daily ultrasound and serum estradiol and LH level evaluation will be performed when the mean diameter of the dominant follicle of ≥14 mm. LH surge initiation is defined as a concentration of 180% above the latest serum value available in that patient with a continued rise thereafter to a level of 20 IU/l or more detected by the ECLIA method (Roche Cobas® E 801, Roche Diagnostics, Germany). Embryo transfer will be scheduled by the time of the initiation of LH and embryo stages.

modified Natural protocol The first ultrasound scan will be performed on the second to the fourth day of the menstrual cycle to identify any problem related to the patient's uterus or adnexa. A second ultrasound scan will be performed on the sixth day of the cycle; if there is at least one follicle with a diameter of ≥12 mm, an ultrasound scan will be performed daily. When the dominant follicle's mean diameter is ≥16 mm, human chorionic gonadotropin - hCG (Ovitrelle® 250 μg; Merck, Kenilworth, NJ, USA) will be injected to trigger ovulation. Embryo transfer will be scheduled by the time of the hCG injection and embryo stages.

Serum progesterone level was also evaluated using the electrochemiluminescence immunoassay (Elecssys Progesterone III, Cobas®, Roche diagnosis, Germany) with a CV of 5.2%.

Serum progesterone was measured at 3 time points:

* 1st sample: On day 2 to day 4 of the cycle, before starting the endometrial preparation regime
* 2nd sample:

  * For AC protocol: Before administration of vaginal progesterone
  * For mNC protocol: Before hCG administration
  * For NC protocol: When an LH surge initiation was recorded, i.e., serum LH measured 20 IU/L or more
* 3rd sample: On the day of frozen embryo transfer at 8 a.m. Cycle cancellation

  * Artificial protocol: When the endometrial thickness is below 7mm after a duration of estradiol administration of ≥21 days or the emergence of a dominant follicle.
  * Natural cycle protocol: When there is no development of follicle, or no dominant follicle (≥14 mm), or no onset of LH surge observed after a duration of ≥21 days or unexpected spontaneous ovulation appears.
  * modified Natural cycle protocol: When there is no developing follicle (>16mm) observed after a duration of ≥21 days or pre-hCG unexpected spontaneous ovulation appears.
  * Both protocols: When there is no embryo surviving after thawing.

Frozen embryo transfer:

A maximum of 2 day-3 and one day-5 embryos will be thawed on the day of embryo transfer, three days after the start of progesterone. Two hours after thawing, surviving embryos will be transferred into the uterus under ultrasound guidance using a soft uterine catheter (Gynétics®, Belgium).

A series of progesterone levels evaluation will be performed at three times: (1) at the start of the cycle, (2) Before the time the embryo transfer is scheduled, (3) On the day of embryo transfer.

The blood sample at the start of the cycle will be stored for further epigenetics analysis.

Future babies' health will also be performed separately.

ELIGIBILITY:
Inclusion Criteria:

* Aged of 18 to 45
* Having menstrual cycle duration of 24 to 38 days
* Undergoing no more than 3 previous IVF/ICSI - FET cycles
* Planning a frozen-thawed embryo transfer
* Agreeing to have no more than 2 day 3 and 1 day 5 embryos transferred
* Not participating in another IVF study at the same time

Exclusion Criteria:

* Menopausal/ Anovulatory women
* Having contraindication for exogenous hormones administration: breast cancer, risks of venous thromboembolism
* Having embryos from in vitro Maturation or oocyte donation or PGT (pre-implantation genetics testings) cycles
* Having uterine abnormalities (e.g., adenomyosis, intrauterine adhesions, unicornuate/ bicornuate/ arcuate uterus; unremoved hydrosalpinx, endometrial polyp)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1428 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Live birth rate after one frozen embryo transfer cycle | At 24 weeks of gestation
  Live birth is defined as the complete expulsion or extraction from a woman of a product of fertilisation, after 24 completed weeks of gestational age; which, after such separation, breathes or shows any other evidence of life, such as heart beat, umbilical cord pulsation or definite movement of voluntary muscles, irrespective of whether the umbilical cord has been cut or the placenta is attached. A birth weight of 350 grams or more can be used if gestational age is unknown (twins are a single count).

SECONDARY OUTCOMES:
Positive pregnancy test | At 2 weeks after embryo placement
  Serum ß-hCG ≥25mIU/mL
Clinical pregnancy | At 5 weeks after embryo placement
  Having at least one gestational sac on ultrasound at 7 weeks' gestation with the detection of heart beat activity
Ongoing pregnancy | At 10 weeks after embryo placement
  Having at least 1 gestational sac on ultrasound at 12 weeks' gestation with heart beat activity
Implantation | At 3 weeks after embryo placement
  Implantation rate is explained as the number of gestational sacs per number of embryos transferred.
Ectopic pregnancy | At 12 weeks of gestation
  A pregnancy outside the uterine cavity, diagnosed by ultrasound, surgical visualisation, or histopathology
Miscarriage | At 20 weeks of gestation
  The spontaneous loss of an intra-uterine pregnancy prior to or at 20 completed weeks of gestational age
Preterm delivery | At 22, 28, 32 weeks and 37 weeks of gestation
  Multiple definitions, defined as delivery at <24, <28, <32, <37 completed weeks
Endometrial preparation cycles cancelation | At 3 weeks from the start of treatment cycle
  Cycle cancelling due to:
  * Artificial protocol: When the endometrial thickness is below 7mm after a duration of estradiol administration of ≥21 days or the emergence of a dominant follicle.
  * Natural cycle protocol: When there is no development of follicle, or no dominant follicle (≥14 mm), or no onset of LH surge observed after a duration of ≥21 days or unexpected spontaneous ovulation appears.
  * modified Natural cycle protocol: When there is no developing follicle (>16mm) observed after a duration of ≥21 days or pre-hCG unexpected spontaneous ovulation appears.
  * Both protocols: When there is no embryo surviving after thawing.
  * Fluid in uterine cavity
  * Side effects of taking exogenous hormones: severe migraine/headache, mood swings, vaginal bleeding, nausea; venous thromboembolism, stroke.
  * Patient preferences
Gestational diabetes mellitus | At 24 to 28 weeks of gestation
  using a 75g oral glucose tolerance test
Hypertensive disorders of pregnancy | At 20 weeks of gestation or beyond
  Pregnancy-induced hypertension, pre-eclampsia and eclampsia
Birth weight | At the time of delivery
  Weight of singletons and twins
Low birth weight | At birth
  Weight < 2500 gm at birth
Very low birth weight | At birth
  Weight < 1500 gm at birth
High birth weight | At birth
  Weight >4000 gm at birth
Very high birth weight | At birth
  Weight >4500 gm at birth
Major congenital abnormalities | At birth
  Structural, functional, and genetic anomalies, that occur during pregnancy, and identified antenatally, at birth, or later in life, and require surgical repair of a defect, or are visually evident, or are life-threatening, or cause death. Any congenital anomaly will be included as followed definition of congenital abnormalities in Surveillance of Congenital Anomalies by Division of Birth Defects and Developmental Disabilities, NCBDDD, Centers for Disease Control and Prevention (2020).
Admission to NICU | At birth
  The admittance of the newborn to NICU
Venous thromboembolism relating to medication | From the start of treatment up to 10 weeks of gestation
  Venous thromboembolism is diagnosed after clinical examination, ultrasound scan and blood test
Multiple pregnancy | At 6 to 8 weeks' gestation
  ≥1 gestational sac at early pregnancy ultrasound
Multiple delivery | At 24 weeks' gestation
  Birth of more than one baby beyond 24 weeks
Cost-effectiveness | Two year after randomization
  Including direct and indirect costs; costs related to complications treatment. Cost data will be collected for a supplementary analysis and will be reported in a separated paper.
Still birth | At 20 weeks' gestation
  The death of a fetus prior to the complete expulsion or extraction from its mother after 20 completed weeks of gestational age. The death is determined by the fact that, after such separation, the fetus does not breathe or show any other evidence of life, such as heartbeat, umbilical cord pulsation, or definite movement of voluntary muscles.

CONTACTS AND LOCATIONS:
Overall Officials: Lan N Vuong, MD, PhD, Principal Investigator — University of Medicine and Pharmacy at Ho Chi Minh City
Locations (1):
- My Duc Hospital, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ho VNA, Pham TD, Nguyen NT, Wang R, Norman RJ, Mol BW, Ho TM, Vuong LN. Livebirth rate after one frozen embryo transfer in ovulatory women starting with natural, modified natural, or artificial endometrial preparation in Viet Nam: an open-label randomised controlled trial. Lancet. 2024 Jul 20;404(10449):266-275. doi: 10.1016/S0140-6736(24)00756-6. Epub 2024 Jun 26. PMID 38944045